CLINICAL TRIAL: NCT06246643
Title: A Single Arm, Open-label, Multicenter Phase 2 Study of Regorafenib in Participants Who Have Been Treated in a Previous Bayer-sponsored Regorafenib Study (Monotherapy or Combination Treatment) That Has Reached the Primary Completion Endpoint or the Main Data Analysis or Has Been Stopped Prematurely.
Brief Title: A Study of Continued Treatment With Regorafenib in Participants With Solid Tumors Who Have Participated in Other Bayer Studies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22551; 2023-507084-19-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-01-14; First posted 2024-02-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Solid Malignant Tumors
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental): Adult and pediatric patients from completed Bayer-sponsored regorafenib trials who are benefiting from regorafenib treatment.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Participants will be treated with the regorafenib dose taken during the last cycle of the feeder study. Adult participants will receive either 60, 80, 90, 120, or 160 mg orally (p.o.) once daily (qd) for 3 weeks of every 4-week cycle (i.e. 3 weeks on, 1 week off). Pediatric participants will receive 82 mg/m^2 p.o. qd for 14 days, in a 14 days on/7 days off schedule (21-day cycle).

SUMMARY:
Regorafenib is an anti-cancer drug that blocks several proteins which are involved in the growth of cancer. It has been approved for different types of cancers of the digestive system and is being tested for use in some other solid tumors. Cancers that start in an organ, a muscle, or a bone form a solid tumor.

This study is for participants with solid tumors who have been taking regorafenib in other Bayer studies. They can continue taking regorafenib if it is working when treatment with regorafenib in their previous study ends.

The main purpose of this study is to find:

* How safe is the continued treatment with regorafenib in participants with solid tumors?
* How well is the continued treatment with regorafenib tolerated by participants with solid tumors?

Participants will continue with the same dose of regorafenib that they were taking in their previous study as long as the treatment works for them/they want to continue the treatment/other medical conditions do not prevent them from participating in the study. For participants that are under 18 years of age, regorafenib tablets will be taken by mouth once daily for 2 weeks and repeat again after a 1-week gap. For participants that are over 18 years of age, regorafenib tablets will be taken by mouth once daily for 3 weeks and repeat again after a 1-week gap.

At the start of the study, researchers will review participants' records from the previous study. During the study, researchers will use blood samples and X-rays taken from participants under the age of 18 years to check how safe regorafenib is for children. They will also monitor any medical problems that participants may have during the study. After the last dose, follow-up will be done either within 14 days when participants visit their study doctor or within 30-35 days by phone call.

Both the researchers and the participants will know the dose of regorafenib the participants receive during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently participating in any Bayer-sponsored regorafenib study and is receiving regorafenib as study treatment.
* Participant is currently benefiting from treatment with regorafenib monotherapy. All participants must meet criteria to initiate a subsequent cycle of therapy, as determined by the guidelines of the feeder protocol.
* Any ongoing adverse events that require temporary treatment interruption must be resolved to baseline grade or assessed as stable and not requiring further treatment interruption by the investigator.

Exclusion Criteria:

* Ineligibility, for medical reasons, to start the subsequent cycle in the respective feeder study.
* Participants with a beta-human chorionic gonadotropin (hCG) test result consistent with pregnancy.
* Participants are using one or more of the prohibited medications listed in the respective feeder study protocol.
* Participant has been previously permanently discontinued from regorafenib treatment.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2028-04-27 (Estimated); Study Completion 2028-04-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAEs) and protocol-specified AEs and their severity | through study completion, an average of 2.5 year

SECONDARY OUTCOMES:
Number of participants with dose modifications | through study completion, an average of 2.5 year

CONTACTS AND LOCATIONS:
Locations (7):
- France (3):
  - Hôpital Beaujon - Clichy, Clichy
  - Hopital Claude Huriez - Lille, Lille
  - Hôpital Paul Brousse - Villejuif, Villejuif
- Saitama Cancer Center, Kitaadachi-gun, Saitama, Japan
- Seoul National University Hospital, Seoul, Seoul Teugbyeolsi, South Korea
- Hospital Infantil Universitario Nino Jesus | Oncologia Pediatrica, Madrid, Spain
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22551